CLINICAL TRIAL: NCT05828836
Title: the Impact of Allopurinol of HRQOL in Cirrhotic Patients
Brief Title: Allopurinol and Quality of Life in Liver Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Ahmed Mhrose Glal, assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AqOL
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- allopurinol (Active Comparator)
  Interventions: Drug: Allopurinol Tablet

INTERVENTIONS:
Drug: Allopurinol Tablet — allopurinol300mg once daily
  Arms: allopurinol
Drug: Placebo — placebo once daily
  Arms: placebo

SUMMARY:
The study aims to evaluate the impact of allopurinol on patients' related quality of life.

DETAILED DESCRIPTION:
Cirrhosis is the late stage of liver damage and possess two phases:. The shift from compensated to decompensated cirrhosis is characterized by the onset of complications) which are associated with substantial morbidity and negative Impact on quality of life (QOL)Cirrhosis and its complications have a substantial economic, social, and personal impact on affected patients, as well as their families and caregivers

ELIGIBILITY:
Inclusion Criteria:

cirrhosis adult both sex

Exclusion Criteria:

* renal insufficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Chronic liver disease questionnaire | 6 months
  effect on Chronic liver disease questionnaire score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Tanta, Egypt